CLINICAL TRIAL: NCT02002624
Title: RCT Multicenter Comparison of Patient-Specific Versus Conventional Instrumentation in Primary TKA
Brief Title: Patient-Specific Versus Conventional Instrumentation in TKA
Acronym: Visio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochin Hospital (Ambiguous)
Responsible Party: Principal Investigator, Moussa Hamadouche, MD, PhD, Cochin Hospital
Organization: Cochin Hospital, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCP SC 2837
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Active Comparator): Conventional instrumentation
  Interventions: Device: Conventional instrumentation
- PSI (Experimental): Patient specific instrumentation
  Interventions: Device: PSI

INTERVENTIONS:
Device: PSI
  Other Names: Patient specific instrumentation
  Arms: PSI
Device: Conventional instrumentation
  Arms: Conventional

SUMMARY:
The aim of this prospective multicenter randomized clinical trial (RCT) is to compare the clinical and radiologic results of primary total knee arthroplasty (TKA) using patient-specific versus conventional instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary or secondary osteoarthritis of the knee requiring total knee arthroplasty
* aged between 18 and 85 years
* able to understand information
* affiliated to social security.

Exclusion Criteria:

* active or suspected sepsis
* tumor around the knee
* previous partial or total knee replacement
* presence of hardware that could artifact MRI
* contraindication to MRI
* extra-articular deformation requiring osteotomy around the knee in conjunction with TKA
* social situation that could impair follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mechanical axis | 3 months
  Lower limb mechanical axis was measured on a bipodal standing leg-length anteroposterior radiograph with the patella oriented straight made three months postoperatively, using Roman software version 1.70 (Oswestry, United Kingdom). Postoperative lower limb mechanical axis was calculated from the HKA (hip-knee-ankle) angle between the femoral and tibial mechanical axes, respectively. An HKA angle greater than 180° was indicative of valgus, whereas values lower than 180° indicated varus.

SECONDARY OUTCOMES:
Components position | 3 months
  Also, components position in the coronal plane was measured on both the tibial and femoral sides by the femoral (F) angle between the tangent line of the distal prosthetic condyles and the mechanical axis of the femur, and by the tibial (T) angle between the tangent line of the prosthetic tibial baseplate and the mechanical axis of the tibia. In addition in the sagittal plane, tibial slope (TS) was measured by the angle between the tangent of the tibial baseplate and the posterior cortex of the tibia on a lateral view of the knee made at three-month follow-up.

OTHER OUTCOMES:
Blood loss | 5 days
  According to Mercuriali et al.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Boisgard, MD, PhD, Study Director — University Hospital, Clermont-Ferrand